CLINICAL TRIAL: NCT04967378
Title: Feasibility, Acceptability, and Preliminary Efficacy Study of a Cognitive-Emotional Intervention Program for Homebound Older Adults With Mild Cognitive Impairment
Brief Title: Homebound Elderly People Psychotherapeutic Intervention
Acronym: HEPPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Collaborators: Foundation for Science and Technology, Portugal (Other)
Responsible Party: Principal Investigator, Andreia Jesus, Integrated non-PhD member, University of Coimbra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HEPPI-CINEICC; SFRH/BD/146170/2019 (Other Grant/Funding Number: Foundation for Science and Technology (FCT))
Record Dates: First submitted 2021-06-19; First posted 2021-07-19 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Mild Cognitive Impairment; Depressive Symptoms; Anxiety State
Keywords: Homebound Older Adults; Mild Cognitive Impairment; Depressive and Anxious Symptomatology; Cognitive-Emotional Intervention Program
MeSH Terms: conditions — Cognitive Dysfunction; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEPPI program (Experimental)
  Interventions: Behavioral: HEPPI
- Waiting-list control group (No Intervention): Receives access to HEPPI program at the end of the study.

INTERVENTIONS:
Behavioral: HEPPI — 10 weekly individual sessions, 90 minutes each, at the participants' homes. The content of sessions includes psychoeducation, cognitive training, psychotherapeutic intervention, and compensatory strategy training.
  Other Names: Homebound Elderly People Psychotherapeutic Intervention
  Arms: HEPPI program

SUMMARY:
This study aims to develop, implement, and assess the feasibility, acceptability, and preliminary efficacy of a 10-week structured and individualized cognitive-emotional intervention program for homebound older adults with Mild Cognitive Impairment (MCI) and with depressive and/or anxiety symptoms. Homebound Elderly People Psychotherapeutic Intervention (HEPPI) is designed to maintain or improve memory functioning, reduce depressive and/or anxiety symptoms, and help participants to compensate or adapt to impaired cognitive performance, improving their quality of life and their subjective perception of memory and health.

DETAILED DESCRIPTION:
There is currently a significant increase in the number of homebound older adults due to multiple physical, psychological, and/or social vulnerabilities, who require in-home support services. A substantial proportion of these elderly people has MCI - more specifically amnesic MCI (aMCI) - often associated with depressive and/or anxious symptomatology. Although the general cognitive functioning and the daily functional capacity is relatively preserved, the cognitive impairment and the emotional difficulties have a significant negative impact in their quality of life.

MCI is a pathological risk condition to develop dementia, more specifically Alzheirmer's disease. Thus, a significant part of homebound older adults is in the prodromal phase of this disease, which represents a key moment for its early detection and for the application of appropriate interventions. Indeed, older adults are able to learn new information and memory strategies, as well as adapt their behavior, allowing them to benefit from such interventions.

The intervention programs focusing on cognition and MCI related symptomatology have revealed to maintain or improve the mnesic abilities and attention capacity in older people, as well as reduce depressive and/or anxiety symptoms. However, despite the growing research, there are few studies applying and assessing the effectiveness of these programs in homebound older adults. Therefore, the purpose of this study is to examine the feasibility, acceptability, and preliminary efficacy of the HEPPI program - a cognitive-emotional intervention program for homebound older adults with Mild Cognitive Impairment and with depressive and/or anxiety symptoms.

A sample of homebound older adults over 65 years old with aMCI and with depressive and/or anxiety symptoms is being recruited through contact with national entities that identify and work directly with this population, and through contact with their social support network. Participants who demonstrate interest are informed about the aims and procedures of the study, and asked to sign an informed consent form before eligibility assessment. Eligible participants are randomly assigned to either an experimental group, who receive the intervention, or a waiting-list control group, who will receive access to HEPPI program at the end of the study. Both groups complete a neuropsychological protocol to assess measures of cognition, psychological health, subjective memory complaints, quality of life, personality, and functional capacity. This protocol is applied in two different moments: at baseline (PRE) and one week after the intervention (POS1). The study procedures take place at the participants' homes.

ELIGIBILITY:
Inclusion Criteria:

* Homebound older adults over 65 years old;
* Presence of aMCI;
* Presence of depressive and/or anxiety symptoms;
* Residence in mainland Portugal;
* Provision of written informed consent by participants.

Exclusion Criteria:

* Presence of a dementia diagnosis;
* Presence or history of other significant neurological conditions;
* Presence of severe psychiatric illnesses;
* Presence of comorbid medical conditions associated with cognition decline;
* Use of psychotropic medication;
* Presence of alcoholism or toxicomania;
* Significant impairment of vision, hearing, communication or manual dexterity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of HEPPI program | Baseline
  Measured by recruitment rate
Feasibility of HEPPI program | Immediately after the intervention
  Measured by drop-out rate
Acceptability of HEPPI program | 1 week after the intervention
  Assessed with a questionnaire that includes questions regarding the participants' satisfaction with the program, their intention to use the program, the usefulness and relevance of the program, and its demandingness.

SECONDARY OUTCOMES:
Changes in General Cognitive Function | Baseline, 1 week after the intervention
  Measured by Addenbrooke's Cognitive Examination-Revised (ACE-R) - Higher scores indicate a better outcome
Changes in Verbal Memory | Baseline, 1 week after the intervention
  Measured by Word List I and II (WMS-III) - Higher scores indicate a better outcome
Changes in Episodic Memory | Baseline, 1 week after the intervention
  Measured by Logical Memory I and II (WMS-III) - Higher scores indicate a better outcome
Changes in Sustained Attention | Baseline, 1 week after the intervention
  Measured by Coding-Digit Symbol (WAIS-III) - Higher scores indicate a better outcome
Changes in Depressive Symptomatology | Baseline, 1 week after the intervention
  Measured by Geriatric Depression Scale-30 (GDS-30) - Lower scores indicate a better outcome
Changes in Anxious Symptomatology | Baseline, 1 week after the intervention
  Measured by Geriatric Anxiety Inventory (GAI) - Lower scores indicate a better outcome
Changes in Subjective Memory Complaints | Baseline, 1 week after the intervention
  Measured by Subjective Memory Complaints Scale (QSM) - Lower scores indicate a better outcome
Changes in Quality of Life | Baseline, 1 week after the intervention
  Measured by World Health Organization Quality of Life-OLD Module (WHOQOL-OLD) - Higher scores indicate a better outcome
Changes in Functional Capacity | Baseline, 1 week after the intervention
  Measured by Adults and Older Adults Functional Assessment Inventory (IAFAI) - Lower scores indicate a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Research in Neuropsychology and Cognitive Behavioral Intervention (CINEICC), Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No